CLINICAL TRIAL: NCT03762876
Title: Evaluation of Trans-Hepatic Flow Changes in Major Hepatectomy-THEFLOW Study
Brief Title: Evaluation of Trans-Hepatic Flow Changes in Major Hepatectomy
Acronym: THEFLOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. A. Mehrabi, Professsor, Head of the Division of Liver Surgery and Visceral Transplantation, University Hospital Heidelberg
Other Study IDs: S-576/2017
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Major Hepatectomy
Keywords: Hepatectomy; Trans-hepatic flow; Post-hepatectomy liver failure; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Changes in trans-hepatic flow after major and extended hepatectomy (EH) can lead to small for size and flow syndrome (SFSF), which is associated with a significantly higher rate of morbidity and mortality. The current therapies for SFSF are not effective because tissue damage following SFSF is usually irreversible and the liver parenchyma loses the ability to regenerate. Therefore, the best approach to improve patient survival is to predict SFSF and perform adequate intraoperative preventive procedures.

Portal vein flow (PVF), hepatic artery flow (HAF), and portal vein pressure (PVP) are the main criteria for development of SFSF after living donor liver transplantation. The mechanisms that change trans-hepatic flow are similar after hepatectomy and living donor liver transplantation. Trans-hepatic flow is routinely measured during liver resection, but the effect of these changes on SFSF has not been studied. Identifying the factors that alter trans-hepatic flow after hepatectomy would allow hepatic inflow to be modulated before and after surgery, to prevent SFSF.

Trans-hepatic flow and pressure parameters (PVF, HAF, and PVP) are routinely measured and monitored during liver resection. The aim of the proposed study is to analyze changes in these parameters after major hepatectomy and determine the factors that alter trans-hepatic flow after hepatectomy.

DETAILED DESCRIPTION:
Liver resection is an efficient treatment for primary and secondary hepatic tumors and increases long term survival. Improvements in patient selection criteria, surgical methods, and postoperative care have increased the indications for major and extended hepatectomy (EH). Post-hepatectomy liver failure (PHLF) is a major complication following EH and is called small for size and flow syndrome (SFSF). SFSF significantly increases morbidity and mortality. The current SFSF treatments are not effective because tissue damage following SFSF is irreversible and the liver parenchyma loses the ability to regenerate. The best approach to improve patient survival is to predict SFSF and perform adequate preventive procedures during liver resection. SFSF is caused by changes in trans-hepatic flow and a low future liver remnant volume. Portal vein flow (PVF), hepatic artery flow (HAF), and portal vein pressure (PVP) are the main criteria for SFSF development. Following EH, the ratio of HAF to the remnant liver weight (HAF/100gr) decreases, while the PVF/100gr and the PVP increase. This has various pathologic consequences, which lead to SFSF. Troisi et al. suggested an upper limit of 250 ml/min/100g for PVF to prevent SFSF after living donor liver transplantation. A vascular modulation that decreases the PVF/100gr and PVP and increases the HAF/100gr may prevent SFSF. The mechanisms that alter trans-hepatic flow after hepatectomy and living donor transplantation are similar, but the effect of these changes on SFSF has not been studied following liver resection. Exploring the changes in trans-hepatic flow after major and extended hepatectomy and determining the factors that influence these changes would allow us to modulate hepatic inflow during hepatectomy to prevent PHLF.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Undergoing major or central liver resection
* Aged above 18 years

Exclusion Criteria:

* Cirrhosis
* Previous surgery of the hepatoduodenal ligament
* Status after transjugular intrahepatic portosystemic shunt
* Metabolic liver diseases
* Cardiac failure
* Pulmonary hypertension
* Portal vein thrombosis
* Portal vein hypertension
* Vascular malformation
* Not able to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent Major hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Portal vein flow | One day

SECONDARY OUTCOMES:
Portal vein pressure | One day
  Vein pressure (mmHg)
Hepatic artery flow | One day
Central vein pressure | One day
  Vein pressure (mmHg)
Mean arterial pressure | One day
Post-hepatectomy liver failure | Three months
  Based on the ISGLS criteria
Rate of morbidity | Three months
  Based on the Clavien-Dindo classification
Rate of mortality | Three months
  All cause death events
Grade of liver stiffness | Three months
  Via fibroscan before and after resection

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Golriz, MD, Principal Investigator — Department of General, Visceral and Transplant Surgery, University Hospital; Arianeb Mehrabi, MD, Study Director — Department of General, Visceral and Transplant Surgery, University Hospital
Locations (1):
- Division of Visceral Transplantation, Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Golriz M, Lemekhova A, Khajeh E, Ghamarnejad O, Al-Saeedi M, Strobel O, Hackert T, Muller-Stich B, Schneider M, Berchtold C, Tinoush P, Mayer P, Chang DH, Weiss KH, Hoffmann K, Mehrabi A. Evaluation of the role of transhepatic flow in postoperative outcomes following major hepatectomy (THEFLOW): study protocol for a single-centre, non-interventional cohort study. BMJ Open. 2019 Oct 11;9(10):e029618. doi: 10.1136/bmjopen-2019-029618. PMID 31604785